CLINICAL TRIAL: NCT01110655
Title: Incidence and Cause of Hyponatremia in Endurance Runners, Also to Determine if Oral Hypertonic Saline is as Efficacious as Intravenous Hypertonic Saline in the Correction of Below Normal Blood Sodium Concentrations in Runners With Hyponatremia Without Neurological Symptoms
Brief Title: The Efficacy of Oral Versus Intravenous Hypertonic Saline Administration in Runners With Exercise-Associated Hyponatremia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western States Endurance Run Research Foundation (Other)
Responsible Party: Martin D. Hoffman, MD, Western States Endurance Run
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WSER 2009
Record Dates: First submitted 2010-04-23; First posted 2010-04-26 (Estimated); Last update posted 2010-04-26 (Estimated); Status verified 2010-04

CONDITIONS: Exercise-associated Hyponatremia
Keywords: Exercise-associated hyponatremia; Randomized treatment trial; Endurance runners
MeSH Terms: interventions — Saline Solution, Hypertonic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous hypertonic saline (Experimental)
  Interventions: Other: Intravenous hypertonic Saline
- Oral hypertonic saline (Experimental)
  Interventions: Other: Oral hypertonic saline

INTERVENTIONS:
Other: Intravenous hypertonic Saline — Intravenous 100mL bolus of 3% saline
  Arms: Intravenous hypertonic saline
Other: Oral hypertonic saline — Oral 100mL bolus of 3% saline
  Arms: Oral hypertonic saline

SUMMARY:
The purpose of the study is to 1) evaluate incidence and primary cause of exercise-associated Hyponatremia (EAH) in race finishers participating in the Western States 100-mile Endurance Run, 2) determine if the ingestion of oral hypertonic saline (high salt) is as effective as intravenous administration of hypertonic saline to elevate below-normal blood salt concentrations (EAH) at the end of the Western States Endurance Run, and 3) determine if oral and intravenous hypertonic saline solutions are equally as effective at reversing mild (without altered mental status) symptoms associated with EAH.

ELIGIBILITY:
Inclusion Criteria:

* consenting Western States 100 race finisher
* hyponatremic

Exclusion Criteria:

* altered mental status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Blood sodium concentration post administration of oral or IV hypertonic saline. | 1 hour post administration of hypertonic saline

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Hoffman, MD, Study Chair — Western States Endurance Run Foundation
Locations (1):
- Western States Endurance Run, Sacramento, California, United States